CLINICAL TRIAL: NCT00298792
Title: Individualized Treatment Program for Alcohol Problems
Acronym: IATP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Mark D. Litt, Ph.D., Principal Investigator, University of Connecticut Health Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIAAALIT014202-02; NIH grant 1 R21 AA14202
Record Dates: First submitted 2006-03-01; First posted 2006-03-03 (Estimated); Last update posted 2009-04-15 (Estimated); Status verified 2009-04

CONDITIONS: Alcohol Dependence
Keywords: Cognitive Behavioral Treatment; Alcohol Dependence; Functional Analysis; Experience Sampling; Interactive Voice Response
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Individualized Assessment & treatment (Experimental): Individualized treatment for alcohol dependent persons, based on momentary assessment of high-risk situations and recorded coping abilities.
  Interventions: Behavioral: Cognitive Behavioral Treatment; Behavioral: Cognitive-behavioral treatment
- Packaged Cognitive-Behavioral Treatment (Active Comparator): Manualized cognitive-behavioral treatment for alcohol dependent persons.
  Interventions: Behavioral: Cognitive Behavioral Treatment; Behavioral: Cognitive-behavioral treatment

INTERVENTIONS:
Behavioral: Cognitive Behavioral Treatment — Psychosocial treatment emphasizing teaching of coping skills to maintain sobriety.
Behavioral: Cognitive-behavioral treatment — Psychosocial treatment emphasizing teaching of coping skills to maintain sobriety

SUMMARY:
The purpose of this study is to determine if a treatment for alcohol dependence that is specifically tailored to patients' patterns of drinking and coping strategies can result in better outcomes than more standardized treatments.

DETAILED DESCRIPTION:
Despite the popularity of Cognitive-Behavioral Treatment (CBT) in substance use disorders, recent findings have indicated that CBT may be no more effective than other, less theoretically driven, treatments, and that CBT treatments often fail to result in coping skills acquisition. In order to explore the possibility that current manual-driven modes of CBT delivery may not be adequate to successfully teach coping skills, we are proposing a pilot project for the development of an individualized assessment and cognitive-behavioral treatment program (IATP) for alcohol-dependent persons, in which experience sampling conducted via random calls to cell-phones is used to provide data to create individualized treatment plans. Data collected during experience sampling will include momentary assessments of patients' cognitions, affects, and coping behaviors with respect to drinking.

Participants will be 112 men and women meeting criteria for alcohol dependence, who will be randomly assigned to either a standard packaged manual-driven cognitive-behavioral treatment program (PCBT) like that used in Project MATCH, or to IATP. Patients in both treatments will be asked to engage in experience sampling for two weeks prior to treatment, and for another two weeks after treatment has ended, in order to compare in-vivo measures of coping skills utilization, pre- and posttreatment, between the two groups. Therapy will be conducted over 12 sessions in both treatments. In IATP, the information gathered from experience sampling will form the basis of a functional analysis of patients' drinking and drinking urges during the monitoring period. Cognitive appraisals, moods and coping responses will be evaluated as antecedents and consequences of drinking behavior. Therapists will use the information to address specific cognitions, affects, and behaviors that are adaptive and maladaptive, and will work with the patient to substitute adaptive coping tactics instead. In PCBT the experience sampling data will not be specifically used in therapy, but will still provide in-vivo measures of drinking and coping skills. It is hypothesized that IATP will yield significantly better coping skills acquisition than will PCBT, and that change in coping skills will predict better posttreatment outcomes for IATP. These results would have implications for our delivery of treatment, and for the validity of coping skills training for alcohol addiction.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients 18 years of age or older.
* Participants will have a current DSM-IV diagnosis of alcohol dependence.
* Participants will have signed a witnessed informed consent.

Exclusion Criteria:

* Participants who meet current DSM-IV criteria for bipolar disorder, schizophrenia, dementia, or a psychological disorder requiring medication.
* Participants who have had more than seven days of inpatient treatment for substance use disorders in the 30 days previous to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2006-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Alcohol consumption | Pre - Post

SECONDARY OUTCOMES:
Alcohol-related life problems | Pre - Post

CONTACTS AND LOCATIONS:
Overall Officials: Mark D. Litt, PhD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States